CLINICAL TRIAL: NCT06298760
Title: The Effect of Foot Reflexology and Knee Massage Applied With Black Cumin Extract Oil on Pain and Fatigue Symptoms in Elderly People With Knee Osteoarthritis
Brief Title: The Effect of Reflexology and Knee Massage With Black Cumin Oil on Pain and Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Ercan Bakır, assoc prof, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: çörekotu refleksoloji
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Black Seed Oil; Foot Reflexology; Knee Massage; Pain; Fatigue; Nursing
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: After randomization, participants were divided into 30 participants in each group.
  were divided into five groups:Groups; It consisted of 1) Reflexology with Black Cumin, 2) Placebo Reflexology, 3) Knee Massage with Black Cumin, 4) Placebo Knee Massage and 5) Control groups. "Patient Information Form", "Kellgren and Lawrence", "Pain Visual Analog Scale (A-VAS)", "Fatigue Severity Scale and Western Ontario and McMaster Universities Osteoarthritis Index "WOMAC" were applied to the participants. Participants in the application groups were administered once a week for 6 weeks. The session lasted 30 minutes. The control group was allowed to continue routine treatment and care without any intervention. Data were collected by applying questionnaires to the participants in the 1st and 6th weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Knee Massage With Black Cumin Oil Group (Experimental): Necessary explanations were made to the patients in this group. Before application, 5 drops of black cumin oil were applied to the patient's knee for 20 minutes. waited. After making sure that there was no allergy, both knees were massaged with oil for a total of 30 minutes.
  Interventions: Combination Product: Knee Massage With Black Cumin Oil Group:
- Placebo Knee Massage Application Group (Placebo Comparator): Patients in this group received a 30-minute knee massage with pure petroleum jelly.
  Interventions: Combination Product: placebo group
- Foot Reflexology Group With Black Cumin Oil (Experimental): Patients in this group underwent foot reflexology with pure black cumin oil for 40 minutes on both feet.
  Interventions: Combination Product: Foot Reflexology Group With Black Cumin Oil
- Placebo Foot Reflexology Group (Placebo Comparator): Patients in this group underwent foot reflexology with vaseline for 40 minutes on both feet.
  Interventions: Combination Product: placebo group
- Control Group (No Intervention): No intervention was performed on patients in this group. Followed for 6 weeks. Face-to-face meetings were held once a week.

INTERVENTIONS:
Combination Product: Knee Massage With Black Cumin Oil Group: — The patients received a knee massage with black cumin oil once a week for approximately 30 minutes for 6 weeks.
  Arms: Knee Massage With Black Cumin Oil Group
Combination Product: Foot Reflexology Group With Black Cumin Oil — The patients underwent foot reflexology with black cumin oil once a week for approximately 40 minutes for 6 weeks.
  Arms: Foot Reflexology Group With Black Cumin Oil
Combination Product: placebo group — Applications were made with vaseline
  Arms: Placebo Foot Reflexology Group; Placebo Knee Massage Application Group

SUMMARY:
In this study, black cumin extract oil was used in elderly individuals with Knee Osteoarthritis (OA). The effects of foot reflexology and knee massage on pain and fatigue symptoms. It is aimed to examine and research which of these two applications is more effective.The study, planned as a randomized controlled experimental study, included a total of 150 participants.

The data consists of participants who receive outpatient treatment in the Physical Therapy and Rehabilitation Unit at a university hospital, are over 65 years old, and have no problems with their perception after the Mini Mental Test. After randomization, participants were divided into five groups, with 30 participants in each group. Groups; It consisted of 1) Reflexology with Black Cumin, 2) Placebo Reflexology, 3) Knee Massage with Black Cumin, 4) Placebo Knee Massage and 5) Control groups.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is an insidiously progressive disease that causes structural destruction in the joints, cartilage tissue and subchondrial bone, inflammation in the synovial tissue and consequently osteophyte formations; It is an irreversible, degenerative joint disease.Its incidence increases with age and it is the second most common disease in 50% of individuals over the age of 65.It is also the most common cause of chronic pain, fatigue, functional disability, physical disability and limitation in individuals in this age group.The primary complaint of patients with knee OA is pain. Pain is usually; It is seen in intraarticular and periarticular regions. Pain is initially intermittent, mild, and limited to the joint area. In the later stages of the disease, the pain is deep, aching and intense.Although patients experience difficulty in their daily living activities due to pain, the main reason why they cannot perform their activities is pain-related fatigue. Although there is no evidence level method to modify the deformations that occur in the joint structure in OA, various treatment methods are available. The primary goal of treatment in individuals with knee OA is to reduce pain, relieve fatigue, prevent deformations and maintain the patients' independence. There are important clinical guidelines for these goals. According to the guidelines in the treatment of osteoarthritis; Classified in 5 Categories: Pharmacological Treatments, Non-Pharmacological Treatments, Intra-artricular Treatments, Surgical Treatments and Complementary and Integrated Treatments (CAM). According to literature reviews, the most frequently used methods by OA patients include aromatherapy, massage and reflexology, and massages generally include black cumin, olive oil, lavender, rosemary, ginger, etc. It is observed that the oils are applied by rubbing them into the knee and these applications reduce pain and fatigue.Black Cumin; The most important active ingredient is thymoquinone (TQ). Thymoquinone is an important component due to its effect on reducing joint inflammation and rheumatic pain, and this feature makes this oil preferred in aromatherapy.Massage; It is defined as a manual work that helps symptom management and control by creating external rhythmic and impulsive pressure on the soft tissues in the body in order to maintain the health of the body and to support healing in case of disease, especially by helping the circulatory system.Reflexology; projection of glands and organs in the body; It corresponds to reflex points on the hands, feet and ears. It is defined as an application aimed at ensuring that body activities are at an optimum level by stimulating these specific points with unique manipulative techniques through the hands. Ease of application of OA patients in addition to standard treatment It will be beneficial for patients to know and use aromatherapy, massage and reflexology methods that will not cause difficulties in terms of accessing and accessing materials.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with knee OA
* Staged according to Kellgren-Lawrence Gonarthrosis staging and Stage 2 and above
* Open to communication and without cognitive problems
* Those aged 65 and over
* Not allergic to the essential oil used
* Those who have no open wounds on their knees or feet and have not undergone any surgery
* VAS- Pain and Fatigue Severity score of 4 and above
* Mini Mental Test (MMT) score >25
* People who agreed to participate in the research were included in the study.

Exclusion Criteria:

* not meeting the inclusion criteria
* Patients who did not agree to participate in the study were not included in the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Pain Score | 6 weeks
  visual analog scale:VAS: It is a scale scored between 0 and 10 points. A score of 0 indicates that the patient has no pain, and a score of 10 indicates that the patient has unbearable pain. The patient gives a score between 0 and 10 depending on the pain condition.

SECONDARY OUTCOMES:
fatigue severity | 6 weeks
  fatigue severity scale (FSS): The scale consists of 9 questions. Each question is scored between 0 and 7. It is a scale that questions the patient's exercise status, motivation, and daily life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bakır, Study Director — erzurum tecnical university
Locations (1):
- Ercan Bakır, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huseini HF, Mohtashami R, Sadeghzadeh E, Shadmanfar S, Hashem-Dabaghian F, Kianbakht S. Efficacy and safety of oral Nigella sativa oil for symptomatic treatment of knee osteoarthritis: A double-blind, randomized, placebo-controlled clinical trial. Complement Ther Clin Pract. 2022 Nov;49:101666. doi: 10.1016/j.ctcp.2022.101666. Epub 2022 Sep 17. PMID 36150238
- [Background] Kooshki A, Forouzan R, Rakhshani MH, Mohammadi M. Effect of Topical Application of Nigella Sativa Oil and Oral Acetaminophen on Pain in Elderly with Knee Osteoarthritis: A Crossover Clinical Trial. Electron Physician. 2016 Nov 25;8(11):3193-3197. doi: 10.19082/3193. eCollection 2016 Nov. PMID 28344755
- [Result] Tuna HI, Babadag B, Ozkaraman A, Balci Alparslan G. Investigation of the effect of black cumin oil on pain in osteoarthritis geriatric individuals. Complement Ther Clin Pract. 2018 May;31:290-294. doi: 10.1016/j.ctcp.2018.03.013. Epub 2018 Mar 22. PMID 29705470